CLINICAL TRIAL: NCT00202865
Title: CANaDian Evaluation of Low DosE Infliximab in Ankylosing Spondylitis
Brief Title: Evaluation of Low Dose Infliximab in Ankylosing Spondylitis (Study P04352)
Acronym: CANDLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04352; 2472
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: infliximab
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: infliximab — Infliximab 3 mg/kg infusions at Weeks 0, 2, and 6 and every 8 weeks thereafter. Subjects who lose response according to a pre-specified criteria at weeks 22 or 38 visit will increase the dose of infliximab to 5 mg/kg (rounded up to the nearest vial).
  Other Names: Remicade; SCH 215596
  Arms: 1
Biological: Placebo — Placebo infusions at Weeks 0, 2, and 6. Subjects will be evaluated at Week 12 after which they will receive infliximab 3 mg/kg at Weeks 16, 18, and 22 then every 8 weeks. Subjects who lose response according to a pre-specified criteria at weeks 22 or 38 visit will increase the dose of infliximab to 5 mg/kg (rounded up to the nearest vial).
  Arms: 2

SUMMARY:
This is a randomized, double-blind, multi-center, placebo-controlled study with two parallel treatment groups (placebo and infliximab) in subjects with ankylosing spondylitis (AS) to evaluate the efficacy of infliximab 3 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Are men or women >=18 years of age at Screening.
* Female subjects of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active during the study) must be using an acceptable method of birth control (eg, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (eg, hysterectomy or tubal ligation), and must continue such precautions for 6 months after receiving the last study agent infusion, and have a negative serum pregnancy test prior to enrollment. Additionally, male subjects who are sexually active, with women of childbearing potential, should ensure that they or their partners are using adequate contraception
* Have had a diagnosis of AS according to the modified 1984 New York criteria, prior to Screening.
* Have active disease, as evidenced by a BASDAI score of >=4 at Baseline and at Screening
* Screening tests must meet the following criteria:

  * Hemoglobin: >=9.0 g/dL (5.6 mmol/L) for men and >=8.5 g/dL (5.3 mmol/L) for women
  * Serum transaminase levels must be within 3 times the ULN
  * Serum creatinine <=1.4 mg/dL (107umol/L).
* Are capable of reading and understanding subject assessment forms and providing written informed consent.
* Have had a documented negative reaction to a PPD skin test (PPD induration < 5 mm) performed within 1 month prior to the first study infusion. If PPD negative, chest x-ray still required.
* Subjects must understand English or French.

Exclusion Criteria:

* Have had a serious infection (eg, sepsis, hepatitis, abscesses, pneumonia, or pyelonephritis), have been hospitalized for an infection, or have been treated with intravenous (IV) antibiotics for an infection within 8 weeks prior to randomization. Less serious infections (eg, acute upper respiratory tract infection, or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
* Have ever had a chronic or recurrent infectious disease including, but not limited to, chronic renal infection, chronic chest infection (eg, bronchiectasis), sinusitis, recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), open, draining, or infected skin wound, or ulcer.
* Have ever had opportunistic infections (eg, herpes zoster (shingles), cytomegalovirus, pneumocystis carinii, aspergillosis, histoplasmosis)
* Have had documented an atypical mycobacteria infection.
* Have had active TB or recent close contact with an individual with active TB or ever had evidence of latent TB.
* Have a chest radiograph (PA and lateral) that displays granulomas or apical fibronodular disease suggestive of previous TB as determined by the investigator.
* Have documented Hepatitis B (surface antigen positive).
* Have documented HIV.
* Have a known malignancy or history of malignancy within 5-year period prior to Screening (with the exception of squamous or basal cell carcinoma of the skin that has been completely excised without evidence of recurrence). Have a history of lymphoproliferative disease including lymphoma, have multiple sclerosis, or other central demyelinating disorder, or have congestive heart failure.
* Have a serious concomitant illness, other than the ones mentioned above, that might interfere with participation in the trial.
* Have a known allergy to murine proteins or other chimeric proteins.
* Have ever received any previous treatment with infliximab, etanercept or other anti-TNF agents prior to first study infusion.
* Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.
* Have a contraindication to any study protocol component.
* Subjects who have a contraindication to the MRI component of the study can be enrolled, however, they will be exempt from all MRI examinations.
* Subjects with unstable doses of NSAIDS, DMARDs, analgesics or corticosteroids at Screening who will continue to receive these medications during the study.
* Subjects who are receiving >10 mg of prednisone (or equivalent) daily.
* Have a documented history of fibromyalgia confirmed by an appropriate physician specialist (ie, rheumatologist).
* Have had a documented history of total ankylosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-01 (Actual)

PRIMARY OUTCOMES:
The proportion of AS assessment responders ASAS20 (ie, a minimum 20% improvement from Baseline according to the ASAS response criteria) at Week 12. | Week 12

SECONDARY OUTCOMES:
Change from Baseline in the magnetic resonance imaging activity score at Week 12. | Week 12
Change from Baseline in BASFI at Week 12 and Week 50. | Week 12 and Week 50
Change from Baseline in BASDAI at Week 12 and Week 50. | Week 12 and Week 50
Change from Baseline in BASGI at Week 12 and Week 50. | Week 12 and Week 50
Change from Baseline in spinal mobility (BASMI) at Week 12 and Week 50. | Week 12 and Week 50
Change from Baseline in spinal mobility (EDASMI) at Week 12 and Week 50. | Week 12 and Week 50
Proportion of subjects achieving an ASAS40 at Week 12 and Week 50. | Week 12 and Week 50
Proportion of subjects achieving an ASAS50 at Week 12 and Week 50. | Week 12 and Week 50
Proportion of subjects achieving an ASAS70 at Week 12 and Week 50. | Week 12 and Week 50
Change from Baseline in the physical component of the SF-36 at Week 12 and Week 50. | Week 12 and Week 50
Assess the treatment survival. | From baseline to week 50
Quantify the number of subjects requiring dose titration. | Week 22 and 38
Assess predictors of response. | Week 12 and 50
Assess predictors of toxicity. | 50 weeks

REFERENCES:
- [Result] Inman RD, Maksymowych WP; CANDLE Study Group. A double-blind, placebo-controlled trial of low dose infliximab in ankylosing spondylitis. J Rheumatol. 2010 Jun;37(6):1203-10. doi: 10.3899/jrheum.091042. Epub 2010 Mar 15. PMID 20231198
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html